CLINICAL TRIAL: NCT03398850
Title: Spontaneous Coronary Artery Dissection anaLysIs of the Brazilian Updated Registry: Epidemiological Data, Clinical Results and Long-Term Follow-up (SCALIBUR Registry).
Brief Title: Spontaneous Coronary Artery Dissection anaLysIs of the Brazilian Updated Registry
Acronym: SCALIBUR
Status: Recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Adriano Caixeta, Professor of Medicine, Hospital Israelita Albert Einstein
Other Study IDs: SCALIBUR Registry
Record Dates: First submitted 2017-12-29; First posted 2018-01-16 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Dissection, Spontaneous
Keywords: spontaneous coronary artery dissection; acute coronary syndrome; coronary angiography; coronary tomography
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective and prospective registry will evaluate demographic and angiographic data in patients with spontaneous coronary artery dissection (SCAD) using medical records, invasive coronary angiography, intravascular imaging and/or computed multislice coronary tomography. The type of treatment applied during index hospitalization (i.e., clinical management, percutaneous coronary intervention or coronary artery bypass grafting) will be evaluated. Long-term follow-up (up to 10 years) will be also reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary manifestations due spontaneous coronary artery dissection
* Angiographic findings of SCAD in coronary angiogram or coronary tomography
* Agreement between two or more invasive cardiologists (adjudicated committee) for the diagnosis.

Exclusion Criteria:

* Non-agreement for SCAD diagnosis
* Coronary dissections due other mechanisms: unstable atherosclerotic plaque or trauma-induced.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The present study population will be selected retrospectively and prospectively from several Brazilian tertiary Hospitals. Clinical data and coronary imaging will be imputed through electronic case report form (eCRF), which will be kept confidential at dedicated server at the Coordinator Center, Hospital Israelita Albert Einstein.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term clinical outcomes in patients presented with spontaneous coronary artery dissection | 10 years
  All major adverse cardiac events will be collected

SECONDARY OUTCOMES:
Multimodality intravascular imaging findings in patients with spontaneous coronary artery dissection. | 10 years
  Multimodality intravascular imaging will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Cade, MD, PhD, Principal Investigator — Hospital Israelita Albert Einstein; Adriano Caixeta, MD, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data from this observational registry will be shared with others researchers and presented at medical conferences.
Supporting Information: Study Protocol, ICF
Time Frame: The first data will be available by 2019
Access Criteria: All researchers will be have the data available upon requested

REFERENCES:
- [Background] Cade J, Mintz GS, Silva RM Filho, Caixeta A. Spontaneous coronary artery dissection and healing documented by optical coherence tomography. Einstein (Sao Paulo). 2016 Jul-Sep;14(3):435-436. doi: 10.1590/S1679-45082016AI3551. Epub 2016 Jul 4. No abstract available. PMID 27383563
- [Background] Cade JR, Abizaid A, Caixeta A. Organized thrombus mimicking spontaneous coronary artery dissection. JACC Cardiovasc Interv. 2014 Dec;7(12):1458. doi: 10.1016/j.jcin.2014.08.004. Epub 2014 Nov 12. No abstract available. PMID 25457056
- [Background] Saw J. Pregnancy-Associated Spontaneous Coronary Artery Dissection Represents an Exceptionally High-Risk Spontaneous Coronary Artery Dissection Cohort. Circ Cardiovasc Interv. 2017 Mar;10(3):e005119. doi: 10.1161/CIRCINTERVENTIONS.117.005119. No abstract available. PMID 28302643
- [Background] Saw J. Coronary angiogram classification of spontaneous coronary artery dissection. Catheter Cardiovasc Interv. 2014 Dec 1;84(7):1115-22. doi: 10.1002/ccd.25293. Epub 2013 Dec 4. PMID 24227590
- [Background] Saw J, Ricci D, Starovoytov A, Fox R, Buller CE. Spontaneous coronary artery dissection: prevalence of predisposing conditions including fibromuscular dysplasia in a tertiary center cohort. JACC Cardiovasc Interv. 2013 Jan;6(1):44-52. doi: 10.1016/j.jcin.2012.08.017. Epub 2012 Dec 19. PMID 23266235
- [Result] Cade JR, Szarf G, de Siqueira ME, Chaves A, Andrea JC, Figueira HR, Gomes MM Jr, Freitas BP, Filgueiras Medeiros J, Dos Santos MR, Fiorotto WB, Daige A, Goncalves R, Cantarelli M, Alves CM, Echenique L, de Brito FS Jr, Perin MA, Born D, Hecht H, Caixeta A. Pregnancy-associated spontaneous coronary artery dissection: insights from a case series of 13 patients. Eur Heart J Cardiovasc Imaging. 2017 Jan;18(1):54-61. doi: 10.1093/ehjci/jew021. Epub 2016 Feb 28. PMID 26928981